CLINICAL TRIAL: NCT07340138
Title: A Phase 1b Study of Pelabresib (DAK539) add-on to Stable Dose of Ruxolitinib in Japanese Adult Patients With Myelofibrosis
Brief Title: Study of Pelabresib add-on to Ruxolitinib in Japanese Adult Patients With Myelofibrosis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDAK539A11101
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Primary Myelofibrosis (PMF); Post-polycythemia Vera Myelofibrosis (Post-PV MF); Post-essential Thrombocythemia Myelofibrosis (Post-ET MF)
Keywords: Pelabresib (DAK539); Ruxolitinib (INC424); Japanese adult participants; Myelofibrosis (MF)
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pelabresib + Ruxolitinib (Experimental): Eligible participants will receive pelabresib 125 mg once daily (QD) in combination with ruxolitinib at doses ranging from 5 to 25 mg twice daily (BID).
  Interventions: Drug: Pelabresib; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Pelabresib — 125 mg orally once daily (QD) on Days 1-14 of each 21-day cycle
  Other Names: DAK539
Drug: Ruxolitinib — 5-25 mg twice daily (BID)
  Other Names: INC424

SUMMARY:
This Phase 1b, multicenter, open-label study aims to evaluate the safety, pharmacokinetics (PK), and preliminary efficacy of pelabresib as add-on to ruxolitinib in Japanese patients with myelofibrosis (MF).

DETAILED DESCRIPTION:
This study consists of three periods: screening, treatment, and follow-up. After a screening period of up to 28 days, between three and nine eligible and evaluable participants will be enrolled to receive pelabresib in addition to a stable dose of ruxolitinib.

The follow-up phase includes a 30-day safety follow-up and a long-term follow-up. Pelabresib will be administered until one of the following occurs: disease progression, unacceptable toxicity, death, participant decision, or investigator decision.

After discontinuation of pelabresib, safety assessments will continue with a safety follow-up visit 30 days after the last dose of pelabresib. Participants will then be contacted for long-term follow-up approximately every 12 weeks after the end of treatment (EOT) for at least three years from the first dose of pelabresib and for at least two years following the last dose of pelabresib, whichever is longer. Long-term follow-up will continue until death, withdrawal from the study, loss to follow-up, or completion of the follow-up period, whichever occurs first.

Safety follow-up and long-term follow-up visits will include assessment for leukemic transformation, which will be conducted throughout the study and for up to two years after treatment. The study will continue until all participants complete long-term follow-up or until access to pelabresib is ensured through a post-trial access program or reimbursement of pelabresib in Japan becomes available.

Japanese safety confirmation will be determined according to the decision rule. The starting dose is 125 milligrams once daily (QD), and no dose escalation or de-escalation for safety confirmation is planned in this study. Initially, three participants will receive 125 milligrams QD of pelabresib as an add-on to ruxolitinib. The dose-limiting toxicity (DLT) evaluation period for Japanese safety confirmation is 21 days (one cycle).

ELIGIBILITY:
Key Inclusion Criteria:

* Participants have diagnosis of primary myelofibrosis (PMF), post-polycythemia vera MF (Post-PV MF) or post-essential thrombocythemia MF (Post-ET MF) according to the International Consensus Classification (ICC) for Myeloid Neoplasms and Acute Leukemias 2022.
* DIPSS risk category intermediate-1, intermediate-2 or high-risk at screening.
* Participants currently treated with ruxolitinib monotherapy AND who are likely to benefit from the addition of pelabresib to ruxolitinib in the opinion of the investigator.
* Receiving ruxolitinib at a stable dose (5 to 25 mg BID) for at least 8 weeks prior to the first dose of pelabresib.
* Palpable spleen (spleen length below left costal margin [LCM] must be recorded) or documented splenomegaly by MRI or CT (image report must be recorded) at screening.
* Platelet count ≥ 100 × 10^9/L in the absence of growth factor support (including thrombopoietin mimetics/agonists) or platelet transfusions 4 weeks prior to the first dose of pelabresib.
* Blasts < 5% in peripheral blood. Assessment of blasts in peripheral blood is mandatory at screening.

Key Exclusion Criteria:

* Prior splenectomy at any time or splenic irradiation in the previous 6 months
* Prior hematopoietic cell transplant or participants anticipated to receive a hematopoietic cell transplant within 24 weeks from the first dose of pelabresib.
* Blasts ≥ 5% in bone marrow if results available at screening or history of accelerated phase or leukemic transformation.
* History of a malignancy (other than MF, PV or ET) except for adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate-specific antigen for ≥ 1 year prior to start of pelabresib, adequately treated Stage 1 or 2 cancer currently in complete remission, or any other cancer that has been in complete remission for ≥ 3 years
* Received any approved or investigational agent for the treatment of MF except ruxolitinib within 14 days of first dose of pelabresib or within 5 half-lives of the approved or investigational agent, whichever is longer.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-05-29 (Estimated); Primary Completion 2027-11-19 (Estimated); Study Completion 2031-03-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | Up to 21 days
  A dose-limiting toxicity (DLT) is defined as any adverse event or abnormal laboratory finding that is not attributable to the underlying disease, disease progression, intercurrent illness or injury, or concomitant medications, occurring within the first 21 days of pelabresib treatment and meeting the protocol-specified criteria. Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0. For Japanese safety confirmation of the 125 mg QD dose, DLTs will be included in the decision-making process.
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | Through study completion, an average of approximately 4 years
  The analysis of adverse events will include categorization by type, frequency, and severity, as graded by the NCI CTCAE version 5.0.

SECONDARY OUTCOMES:
Plasma concentration time profiles of pelabresib | Cycle 1: Days 1/14 (0/Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours post-dose), Days 2/15 (0/Pre-dose (immediately before the next pelabresib administration)). 1 cycle = 21 days.
  Blood samples for pelabresib pharmacokinetics (PK) will be obtained and evaluated to assess single dose and steady-state plasma PK of pelabresib and summarized using descriptive statistics.
Area Under the plasma concentration-time Curve (AUC) of pelabresib | Cycle 1: Days 1/14 (0/Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours post-dose), Days 2/15 (0/Pre-dose (immediately before the next pelabresib administration)). 1 cycle = 21 days.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) and Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) will be listed and summarized using descriptive statistics.
Maximum observed plasma Concentration (Cmax) of pelabresib | Cycle 1: Days 1/14 (0/Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours post-dose), Days 2/15 (0/Pre-dose (immediately before the next pelabresib administration)). 1 cycle = 21 days.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Time to Maximum observed plasma Concentration (Tmax) of pelabresib | Cycle 1: Days 1/14 (0/Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours post-dose), Days 2/15 (0/Pre-dose (immediately before the next pelabresib administration)). 1 cycle = 21 days.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
Absolute change from baseline and percentage change from baseline in spleen volume over time (Week 24 and 48), as measured by MRI (or CT scan). | Baseline, Week 24, Week 48
  Absolute and percentage change from baseline in spleen volume over time (Week 24 and 48) will be summarized using descriptive summary statistics
Absolute change from baseline and percentage change from baseline in Total Symptom Score (TSS) over time (until Week 48), as measured by the Myelofibrosis Symptom Assessment Form (MFSAF) v4.0 | Baseline and up to Week 48
  Absolute change from baseline and percentage change from baseline in Total Symptom Score (TSS) over time (until Week 48) are defined as the difference and percent difference from baseline in TSS at each time point, as measured by the Myelofibrosis Symptom Assessment Form (MFSAF) v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No